CLINICAL TRIAL: NCT05902689
Title: Application of Sticky Bone and Bio-Oss Collagen in Alveolar Ridge Preservation: A Randomized Controlled Clinical Trial
Brief Title: Application of Sticky Bone and Bio-Oss Collagen in Alveolar Ridge Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0369
Record Dates: First submitted 2023-06-01; First posted 2023-06-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-03

CONDITIONS: Alveolar Bone Resorption
Keywords: alveolar ridge preservation; Bio-OSS Collagen; sticky bone

STUDY DESIGN:
Intervention Model Description: The control group underwent natural healing, and the experimental group underwent alveolar ridge preservation using Bio-Oss Collagen and Sticky Bone, respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- blank group (No Intervention): After non-traumatic tooth extraction, the control group will undergo natural healing.
- Bio-Oss Collagen group (Experimental): After non-traumatic tooth extraction, the Bio-Oss Collagen group will use alveolar ridge preservation with bio-oss collagen
  Interventions: Procedure: alveolar ridge preservation with bio-oss collagen
- Sticky Bone group (Experimental): After non-traumatic tooth extraction, the Sticky Bone group will use Sticky Bone for alveolar ridge preservation
  Interventions: Procedure: alveolar ridge preservation with sticky bone

INTERVENTIONS:
Procedure: alveolar ridge preservation with bio-oss collagen — Alveolar ridge preservation with bio-oss collagen is a surgical method that reduces or limits the physiological resorption of alveolar bone after tooth extraction by implanting bio-oss collagen in the socket and covering the biological barrier membrane.
  Arms: Bio-Oss Collagen group
Procedure: alveolar ridge preservation with sticky bone — Alveolar ridge preservation with sticky bone is a surgical method that reduces or limits the physiological resorption of alveolar bone after tooth extraction by implanting sticky bone in the socket and covering the biological barrier membrane.
  Arms: Sticky Bone group

SUMMARY:
In this experiment, after non-traumatic tooth extraction, the blank group underwent natural healing, and the Bio-Oss Collagen underwent alveolar ridge preservation using Bio-Oss Collagen and the Sticky Bone group using Sticky Bone, to verify the application of Bio-Oss Collagen and Sticky Bone in alveolar ridge preservation

DETAILED DESCRIPTION:
Within 6 months after tooth extraction, the remaining alveolar ridge undergoes varying degrees of absorption, resulting in a decrease in horizontal width and vertical height of the alveolar ridge. The three-dimensional size change of the alveolar socket may affect the implantation of later implants and cause aesthetic and functional problems. Alveolar ridge preservation can maintain the volume of the alveolar socket, prevent soft tissue from growing into undesirable positions, slow down the absorption of the alveolar ridge to some extent, promote new bone formation, and maintain the shape of the extraction socket. This is crucial for later implant treatment for missing teeth. In this experiment, after non-traumatic tooth extraction, the blank group underwent natural healing, and the Bio-Oss Collagen group underwent alveolar ridge preservation using Bio-Oss Collagen and the Sticky Bone group using Sticky Bone, respectively, to verify the application of Bio-Oss Collagen and Sticky Bone in alveolar ridge preservation

ELIGIBILITY:
Inclusion Criteria:

1. The presence of one adjacent tooth at the extraction site
2. Adequate oral hygiene (plaque index <20%;bleeding on probing <25% )
3. Need for tooth extraction due to endodontic，periapical or periodontal disease.
4. Presence of ≥ 2 mm of keratinized tissue
5. the extraction sockets have no more than 50% of buccal alveolar bone loss(Integrity of alveolar bone walls)

Exclusion Criteria:

1. Pregnancy or lactation
2. Smoking more than 10 cigarettes per day
3. with no evidence of acute infection such as severe swelling, suppuration at the extraction site
4. Uncontrolled periodontal disease
5. Existence of bone metabolic disease
6. history of malignancy, radiotherapy, or chemotherapy in the past 5 years
7. Administration of bisphosphonates
8. long-term use of NSAIDs
9. Alcohol or drug abuse
10. Infectious disease, such as hepatitis or human immunodeficiency virus (HIV) and/or acquired immunodeficiency syndrome (AIDS)
11. Uncontrolled severe diabetes.( hemoglobin A1c >6.7%)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Changes in horizontal ridge widths | baseline (before the surgery) and six months
  Changes in horizontal ridge widths at 1, 3, and 5 mm below the ridge crest

SECONDARY OUTCOMES:
Changes in the vertical heights of the ridge | baseline (before the surgery) and six months
  Changes in the vertical heights of the ridge at the buccal and lingual crest areas
Thicknesses of the keratinized gingiva | baseline (before the surgery) and six months
  Thicknesses of the keratinized gingiva at 2 and 4mm below the highest point of the gingiva
width of the keratinized gingiva | baseline (before the surgery) and six months
  width of the keratinized gingiva
percentages of newly formed bone | six months
  percentages of newly formed bone and residual bone substitute material in histologic sections
The percentage of residual materials | six months postoperative
The bone density ratio | six months postoperative
The percentage of in alveolar bone volume within the region of interest (ROI) relative to the volume | at baseline
Postoperative response assessed by the Visual Analogue Scale (VAS) questionnaire | 2 weeks post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Li Li Zhou, doctor, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China